CLINICAL TRIAL: NCT00499109
Title: Randomized Phase III Multicenter Trial of RRM1 & ERCC1 Directed Customized Chemotherapy Versus Standard of Care for 1st Line Treatment of Patients With Advanced Non-Small-Cell Lung Cancer
Brief Title: Phase III of RRM1 & ERCC1 Directed Customized Chemotherapy for the Treatment of Patients With NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15005; 105372 (Other: USF IRB); IST 12223 (Other: Sanofi-Aventis US, Inc.); CA129343 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: RRM1; ERCC1; Customized Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Vinorelbine; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E. Dual Agent Chemotherapy (Experimental): Experimental Arm E.
  Patients received treatment according to gene expression strata with four doublet regimens.
  Low ERCC1 and Low RRM1 Group - Gemcitabine (G) and Carboplatin (Cb): GCb Group.
  Low RRM1 and High ERCC1 Group - Gemcitabine (G) and Docetaxel (D): GD Group.
  High RRM1 and Low ERCC1 Group - Docetaxel (D) and Carboplatin (Cb): DCb Group.
  High ERCC1 and High RRM1 Group - Vinorelbine (V) and Docetaxel (D): DV Group.
  Interventions: Drug: Docetaxel; Drug: Vinorelbine; Drug: Carboplatin; Drug: Gemcitabine
- C. Standard of Care Control Arm (Active Comparator): Control Arm C: Gemcitabine and Carboplatin (GCb).
  All patients in arm C were treated with GCb regardless of gene expression levels. Patients received up to 6 cycles, and no maintenance therapy was allowed.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Docetaxel — GD Group: 40 mg/m^2 on days 1 and 8, every 21 days
  DCb Group: 75 mg/m^2 on day 1
  DV Group: 50 mg/m^2 on days 1 and 15, every 28 days
  Other Names: Taxotere
  Arms: E. Dual Agent Chemotherapy
Drug: Vinorelbine — DV Group: 35 mg/m^2 on days 1 and 15
  Other Names: anti-cancer chemotherapy drug
  Arms: E. Dual Agent Chemotherapy
Drug: Carboplatin — GCb Group: Area under the curve (AUC) 5 on day 1, every 21 days
  DCb Group: AUC 6 on day 1, every 21 days
  Control Arm: Patients received up to 6 cycles, and no maintenance therapy was allowed.
  Other Names: Paraplatin
Drug: Gemcitabine — GCb Group: 1,250 mg/m^2 on days 1 and 8
  GD Group: 1,250 mg/m^2 on days 1 and 8
  Control Arm: Patients received up to 6 cycles, and no maintenance therapy was allowed.
  Other Names: Gemzar

SUMMARY:
This is a clinical research study to evaluate if chemotherapy in the experimental arm (E) results in a better outcome compared to patients in the standard of care arm (C).

2:1 randomization to experimental arm (E) or standard arm (C). In arm E, treatment of dual-agent chemotherapy will be selected based on RRM1 and ERCC1 expression at the protein level. In arm C, treatment of dual-agent chemotherapy will be gemcitabine/carboplatin, i.e., standard of care.

DETAILED DESCRIPTION:
Before each cycle, blood tests, vital signs, interim medical history, and a physical exam will be performed. Patients will be carefully checked so that immediate intervention can be initiated should an adverse event (i.e. hypersensitivity) occur.

The last treatment cycle according to the study will be cycle #6, or any earlier cycle. Certain tests will be done within 28 days after the last drug infusion. These include physical exam, vital signs, temperature, weight, adverse event evaluation, imaging studies, and blood work.

The study doctor will see the participants every 6 to 8 weeks for at least 12 months after they start treatment. After that, the participants will be followed every 3 months for an additional 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Non-Small Cell Lung Cancer (NSCLC) of adenocarcinoma, squamous cell carcinoma, large cell carcinoma, or NSCLC not otherwise specified. Patients with suspected NSCLC may enroll prior to the diagnostic biopsy in order to obtain both the diagnostic and molecular analysis-required specimen during the same procedure. Must have blood work within 30 days prior to biopsy to eliminate any unnecessary biopsies on patients that do not qualify (screen failures) due to laboratory values that do not meet the inclusion/exclusion criteria. If a patient has blood work obtained at an outside facility, this can be utilized for the preliminary assessment prior to biopsy, but final inclusion/exclusion values must be obtained within 14 days of start of treatment.
* Willing to undergo biopsy to enable customization of chemotherapy
* Stage IV or IIIB (malignant pleural effusion) NSCLC
* Measurable or evaluable disease by Response Evaluation Criteria In Solid Tumors (RECIST)
* Performance status 0 or 1 by Eastern Cooperative Oncology Group (ECOG) criteria
* Adequate bone marrow function as evidenced by the following (assessed within 14 days of starting treatment): Absolute neutrophil count >= 1,500/mm³, Platelet count >= 100,000/mm³, Hemoglobin >= 8.0 gm/dL
* Prothrombin time (PT) and activated prothrombin time with thromboplastin and kaolin (APTT) within normal laboratory ranges
* Serum creatinine <= 1.5 x upper limit of normal (ULN) assessed within 14 days of starting treatment
* Adequate liver function as evidenced by the following (assessed within 14 days of starting treatment): Total bilirubin must be within normal limits; aspartic transaminase (AST) and alanine transaminase (ALT) <= 2.5 x ULN with a normal alkaline phosphatases; alkaline phosphatases <= 4 x upper limit of normal with normal AST and ALT; patients with elevations of alk phos and AST and/or ALT will be excluded
* Serum calcium <= 1.1 x ULN
* Signed informed consent document
* Women of childbearing potential must have a negative pregnancy test. Men with partners in the childbearing age group and women of childbearing potential must use effective contraception while on treatment and for 6 months thereafter.
* Previous surgery for NSCLC (more that 30 days before study entry)
* Previous radiotherapy (RT) is allowed if: the time between completion of RT and initiation of chemotherapy is at least 7 days; the patient has fully recovered from all toxic effects; at least one target lesion or evaluable disease is outside the radiation field
* Previous chemotherapy allowed if the last dose was administered equal to or greater than 12 months ago. This chemotherapy must have been given in an adjuvant or neoadjuvant mode prior to or after a complete surgical resection (R0 resection) for a NSCLC.
* Patients with stable brain metastases will be allowed to enroll. Stable brain metastases being defined as no progression of brain metastases 28 days after conclusion of definitive treatment as documented by a computed tomography (CT) scan or magnetic resonance imaging (MRI) of the brain. Patients with incidentally discovered asymptomatic brain metastases may be enrolled and treated with chemotherapy without prior brain irradiation if deemed feasible by the treating physician.

Exclusion Criteria:

* Pregnant or lactating
* Prior systemic chemotherapy or immunotherapy for advanced NSCLC.
* Prior malignancies, except: cured non-melanoma skin cancer curatively treated in situ carcinoma of the cervix any other curatively treated malignancy with no evidence of disease recurrence for at least 3 years
* Presence of uncontrolled brain or leptomeningeal metastases
* Peripheral neuropathy or hearing loss of neural origin equal to or greater than grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) v3.0 except if due to trauma
* Other serious illness or medical condition, including but not limited to: congestive heart failure, myocardial infarction within 6 months, significant neurologic or psychiatric disorders that would impact study participation as judged by the treating physician or study chair, infection requiring intravenous (IV) antibiotics, tuberculosis with ongoing therapy at study entry, superior vena cava syndrome (except if controlled with radiation), active peptic ulcer disease, uncontrolled diabetes mellitus as judged by the treating oncologist, any contraindication to high dose corticosteroid therapy (such as herpes simplex, herpes zoster, hepatitis, or other disease)
* Hypercalcemia requiring therapeutic intervention
* Clinically significant ascites and/or pericardial effusion
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* Concurrent treatment with other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2007-05; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Williams, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (9):
- United States (7):
  - Center for Cancer Care & Research/Watson, Lakeland, Florida
  - Leesburg Regional Medical Center, Leesburg, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Johns Hopkins Sidney Kimmell Comprehensive Cancer Center, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Klinik Loewenstein, Löwenstein, Germany
- Ponce School of Medicine, Ponce, Puerto Rico

REFERENCES:
- [Derived] Bepler G, Williams C, Schell MJ, Chen W, Zheng Z, Simon G, Gadgeel S, Zhao X, Schreiber F, Brahmer J, Chiappori A, Tanvetyanon T, Pinder-Schenck M, Gray J, Haura E, Antonia S, Fischer JR. Randomized international phase III trial of ERCC1 and RRM1 expression-based chemotherapy versus gemcitabine/carboplatin in advanced non-small-cell lung cancer. J Clin Oncol. 2013 Jul 1;31(19):2404-12. doi: 10.1200/JCO.2012.46.9783. Epub 2013 May 20. PMID 23690416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were registered onto the trial between May 8, 2007 and December 23, 2010. Study sites included Moffitt Cancer Center and 8 other institutions with locations in the United States, Puerto Rico and Germany.
Period: Overall Study
Arm/Group | E. Dual Agent Chemotherapy | C. Standard of Care Control Arm
Started | 183 | 92
Completed | 165 | 85
Not Completed | 18 | 7

BASELINE CHARACTERISTICS:
Population: All Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | E. Dual Agent Chemotherapy | C. Standard of Care Control Arm | Total
Number analyzed (Participants) | 183 | 92 | 275
Age, Continuous [Mean (Full Range); unit: years] | 64.1 [42.1 to 85] | 62.3 [39.6 to 82.5] | 63.5 [39.6 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 49 | 142
  Male | 90 | 43 | 133
Region of Enrollment [Number; unit: participants]
  United States | 156 | 75 | 231
  Puerto Rico | 3 | 1 | 4
  Germany | 24 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. The data of first documented disease progression or death, as defined by Response Evaluation Criteria In Solid Tumors (RECIST), was recorded, and the time interval from randomization to that date was calculated for each patient and used to generate Kaplan-Meier survival estimates and to calculate the PFS at 6 months.
Time Frame: 6 months
Population: All participants
Measure: Number (95% Confidence Interval); unit: estimated percentage of participants
Arm/Group | E. Dual Agent Chemotherapy | C. Standard of Care Control Arm
Number analyzed (Participants) | 183 | 92
estimated percentage of participants | 52 [45.2 to 59.8] | 56.5 [47.2 to 67.6]

2. Secondary Outcome: Overall Survival (OS)
Description: OS at 12 months, determined from the date of randomization. The time interval from randomization to the date of death was calculated for each patient and used to generate Kaplan-Meier survival estimates and to calculate the overall survival.
Time Frame: 12 months
Population: All participants
Measure: Number (95% Confidence Interval); unit: estimated percentage of participants
Arm/Group | E. Dual Agent Chemotherapy | C. Standard of Care Control Arm
Number analyzed (Participants) | 183 | 92
estimated percentage of participants | 46.1 [39.3 to 54] | 46.6 [37.5 to 58.1]

3. Secondary Outcome: Response Rate (RR)
Description: Number of participants per response category. Response to treatment was determined according to Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 6 months
Population: All evaluable participants
Measure: Number; unit: participants
Arm/Group | E. Dual Agent Chemotherapy | C. Standard of Care Control Arm
Number analyzed (Participants) | 165 | 85
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 64 | 31

ADVERSE EVENTS:
Time Frame: Up to 6 months per participant
Groups:
- Experimental: E1: Docetaxel/Vinorelbine
- Experimental: E2: Docetaxel/Carboplatin
- Experimental: E3: Gemcitabine/Docetaxel
- Experimental: E4; Control: C: Gemcitabine/Carboplatin
Arm/Group | Experimental: E1 | Experimental: E2 | Experimental: E3 | Experimental: E4 | Control: C
Serious Adverse Events (participants affected / at risk) | 21/64 | 12/26 | 16/37 | 20/56 | 32/92
Other Adverse Events (participants affected / at risk) | 57/64 | 24/26 | 34/37 | 54/56 | 86/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: E1 (N=64) | Experimental: E2 (N=26) | Experimental: E3 (N=37) | Experimental: E4 (N=56) | Control: C (N=92)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac General - Other (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constitutional Symptoms - Other (General disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Death not associated with CTCAE term - Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death not associated with CTCAE term - Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 2 (2) | 3 (3) | 8 (10)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Febrile neutropenia: fever - unknown origin W/O clinically or microbiologically documented infection (General disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia) (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hemorrhage, CNS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GI - Abdomen NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/Bleeding - Other (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils/Lung/pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils/Skin/cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils/Wound (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection - Other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Foreign body (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Infection with unknown ANC - Bronchus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC - Wound (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 3 (4)
Neurology - Other (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Obstruction, GU - Ureter (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular/Visual - Other (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain - Abdomen NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain - Back (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain - Bone (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Chest wall (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Chest/thorax NOS (General disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pain - Extremity-limb (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Low Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 4 (5)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence/depressed level of consciousness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (fainting) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular - Other (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 3 (5)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: E1 (N=64) | Experimental: E2 (N=26) | Experimental: E3 (N=37) | Experimental: E4 (N=56) | Control: C (N=92)
Nausea (Gastrointestinal disorders) | 26 (28) | 16 (19) | 13 (17) | 31 (34) | 48 (58)
Constipation (Gastrointestinal disorders) | 18 (19) | 7 (7) | 10 (11) | 17 (18) | 31 (36)
Vomiting (Gastrointestinal disorders) | 17 (22) | 11 (14) | 9 (13) | 13 (13) | 75 (98)
Diarrhea (Gastrointestinal disorders) | 20 (26) | 12 (16) | 13 (29) | 9 (10) | 12 (14)
Anorexia (Gastrointestinal disorders) | 19 (19) | 6 (9) | 10 (15) | 11 (13) | 16 (16)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 14 (14) | 7 (7) | 11 (11) | 7 (7) | 13 (14)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 14 (16) | 0 (0) | 4 (4) | 1 (1) | 4 (4)
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 8 (8) | 3 (3) | 1 (2) | 2 (2) | 3 (3)
Gastrointestinal - Other (Gastrointestinal disorders) | 6 (6) | 2 (6) | 2 (6) | 2 (2) | 4 (4)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 40 (66) | 20 (28) | 28 (37) | 28 (40) | 66 (81)
Fever (in the absence of neutropenia) (General disorders) | 10 (12) | 3 (3) | 9 (12) | 14 (15) | 8 (11)
Insomnia (General disorders) | 10 (10) | 3 (3) | 4 (4) | 7 (7) | 12 (12)
Weight loss (General disorders) | 10 (11) | 1 (3) | 4 (7) | 1 (1) | 10 (13)
Constitutional Symptoms - Other (General disorders) | 6 (10) | 1 (1) | 4 (6) | 3 (7) | 10 (12)
Rigors/chills (General disorders) | 2 (2) | 2 (2) | 1 (1) | 6 (6) | 8 (8)
Sweating (diaphoresis) (General disorders) | 2 (2) | 2 (2) | 2 (2) | 6 (6) | 6 (6)
Pain - Head/headache (General disorders) | 16 (17) | 6 (6) | 5 (5) | 14 (16) | 21 (23)
Pain - Back (General disorders) | 11 (16) | 4 (6) | 5 (5) | 8 (8) | 16 (17)
Pain - Bone (General disorders) | 12 (13) | 1 (1) | 4 (4) | 6 (8) | 8 (9)
Pain - Abdomen NOS (General disorders) | 2 (2) | 2 (3) | 8 (12) | 5 (5) | 10 (11)
Pain - Extremity-limb (General disorders) | 11 (11) | 4 (5) | 3 (4) | 4 (4) | 4 (4)
Pain - Other (General disorders) | 11 (13) | 2 (2) | 4 (4) | 3 (3) | 5 (6)
Pain - Chest/thorax NOS (General disorders) | 5 (6) | 3 (4) | 1 (1) | 5 (6) | 8 (10)
Pain - Joint (General disorders) | 5 (5) | 2 (3) | 2 (2) | 7 (8) | 4 (5)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 32 (32) | 15 (15) | 20 (21) | 12 (12) | 20 (22)
Nail changes (Skin and subcutaneous tissue disorders) | 22 (27) | 4 (4) | 6 (6) | 1 (1) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 (11) | 6 (6) | 6 (6) | 4 (4) | 2 (2)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1) | 2 (2) | 3 (5) | 4 (4)
Neuropathy: sensory (Nervous system disorders) | 25 (33) | 7 (9) | 4 (5) | 11 (11) | 16 (21)
Dizziness (General disorders) | 12 (13) | 4 (5) | 6 (7) | 9 (10) | 19 (21)
Mood alteration - Anxiety (Psychiatric disorders) | 4 (4) | 1 (1) | 2 (2) | 2 (3) | 6 (6)
Low Hemoglobin (Blood and lymphatic system disorders) | 15 (37) | 7 (15) | 4 (8) | 23 (65) | 32 (79)
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (6) | 2 (3) | 3 (3) | 17 (41) | 22 (43)
Low Platelets (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 4 (4) | 20 (40) | 20 (34)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 6 (8) | 11 (13) | 18 (28) | 25 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 5 (5) | 8 (9) | 9 (13) | 22 (25)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (3) | 3 (3) | 4 (4)
Edema: limb (Blood and lymphatic system disorders) | 15 (17) | 4 (5) | 11 (15) | 15 (17) | 15 (18)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 2 (2) | 4 (4) | 4 (5) | 7 (7)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 4 (5) | 3 (3) | 5 (5)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 0 (0) | 2 (3) | 5 (6)
Watery eye (epiphora, tearing) (Eye disorders) | 20 (22) | 3 (3) | 5 (5) | 1 (1) | 2 (2)
Vision-blurred vision (Eye disorders) | 4 (4) | 1 (1) | 4 (4) | 3 (3) | 5 (5)
Dehydration (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (4) | 1 (1) | 3 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Dry mouth/salivary gland (xerostomia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Pain - Throat/pharynx/larynx (General disorders) | 3 (3) | 0 (0) | 0 (0) | 4 (5) | 3 (3)
Pain - Chest wall (General disorders) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Pain - Muscle (General disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 2 (2)
Pain - Oral cavity (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (4)
Mood alteration - Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Cognitive disturbance (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Low Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (10) | 6 (13)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 | 0 (0)
Hemorrhage/Bleeding - Other (General disorders) | 4 (5) | 0 (0) | 3 (4) | 1 (1) | 5 (6)
Febrile neutropenia (Infections and infestations) | 4 (5) | 5 (5) | 0 (0) | 0 (0) | 2 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Infection with unknown ANC - Sinus (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-upper (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 2 (4) | 0 (0) | 7 (12)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (8)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 1 (3)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (4) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (9)
Auditory/Ear - Other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes